CLINICAL TRIAL: NCT01161823
Title: Effect of Nebivolol on Climacteric Disorders in Postmenopausal Women. A Randomized, Open Label Trial
Brief Title: Influence of Nebivolol on Postmenopausal Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Department of Cardiology, Department of Cardiology
Other Study IDs: 451/2009; 2009-011527-31 (EudraCT Number)
Record Dates: First submitted 2010-04-16; First posted 2010-07-14 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2010-04

CONDITIONS: Hot Flashes; Heart Rate; Blood Pressure; Endostatin; Sexual Function
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Nebivolol: 2,5mg or maximum 5mg per day
- Menoflavon: 2 times 1 pill at 40mg Isoflavone per day

SUMMARY:
After menopause the coronary artery disease (CAD) risk increases rapidly to an equivalent risk of men with the same age. The rising incidence of CAD could be a subsequent decline of endogenous estrogen blood levels after the menopause. Estrogen leads to vasodilation and vasoprotection through an increase of Nitric Oxide (NO). NO deficiency results in endothelial stiffness and dysfunction with a subsequent initiation of atherosclerosis. Menopausal status is associated with an increase of the sympathetic nerve activity leading to hypertension, increased heart rate and palpitations. Recent studies show an importance of vasoactive substances (e.g. NO) in the physiology of hot flashes. Thus, hot flashes may be associated with a decreased NO production and release. Additionally, it is well known that during and after menopause women experience a change in sexual function (declined libido and increased dyspareunia) due to decreasing estrogen blood levels. Recently, a new angiostatic parameter - Endostatin (ENST) - has been shown to be involved in EC function. There is also evidence that ENST levels increase during NO stimulation. Nebivolol, a ß-blocker of the third generation, has been shown to release NO to a significant amount in the EC. It is safe and effective in reducing blood pressure to the target level. However, there is no data of the effect of Nebivolol on sexual function, on clinical symptoms (palpitations, increased heart rate and hot flashes) and ENST in postmenopausal women. The present study investigates the effect of a NO-releasing ß-blocker compared to a phytoestrogen therapy considering clinical signs of menopause such as palpitations, hot flashes and sexual functioning in postmenopausal women. Therefore, the use of a ß-blocker treatment is warranted. Further, this study tries to elucidate the role of NO release in postmenopausal symptoms and may gain new insights in the pathophysiology of hot flashes and increased sympathetic nerve activity. Thus, this trial should explore an advantage of Nebivolol therapy in contrast to a phytoestrogen therapy.

Null hypothesis: Climacteric disorders as measured by the MRS-II in patients with a Nebivolol therapy is not lower than in patients with phytoestrogen therapy. Alternative hypothesis: Climacteric disorders in patients as measured by the MRS-II with a Nebivolol therapy is lower than in patients with phytoestrogen therapy.

DETAILED DESCRIPTION:
1. Background

   CAD is the leading cause of mortality for women in US as well as in Austria and most developed countries.

   Major risk factors are hypertension, diabetes and the postmenopausal status. After the menopause the CAD risk increases rapidly to an equivalent risk of men with the same age.

   In all ethnic groups, hypertension is more prevalent among women than men after the age of 59. Over 75 years 75,2 % of females and 63,7% of males perform a hypertensive vascular status.

   Menopausal status is associated with a decline of endogenous estrogen levels resulting in a manifest estrogen deficiency. This estrogen decline is also associated with a subsequent increased risk for CAD.

   The main effect of estrogen is a vasodilatation and an anti-atherosclerotic action through different mechanisms.

   Recent studies are describing that the estrogen deficiency and the subsequently NO deficiency results in a disordered endothelial function and a permanent vasoconstriction, that is one of the major reasons for postmenopausal hypertension and CAD.

   Clinical symptoms of postmenopausal women:

   - Palpitations and tachycardia Postmenopausal women complain about heart palpitations, throbbing and subjective sensed high heart rate and tachycardia, which can be explained by a sympathetic over activity in postmenopausal women.

   This clinical symptoms are associated with a significant decrease in quality of life and well- being in postmenopausal women.

   - Hot flashes Hot flashes are the most common symptom and occur in most postmenopausal women (75%). Hot flashes are experienced as a feeling of intense heat with sweating and rapid heartbeat. The typical duration is between two and thirty minutes. Risk factors for hot flashes are - equal to CVD - high body mass index and smoking.

   Furthermore, it can be supposed that the NO decrease in postmenopausal women is responsible for the hot flashes.

   - Sexuality Sexuality is an important quality-of-life issue, also in elderly. Therefore, sexual dysfunction is considered a serious quality-of-life-related health problem. Furthermore increasing dyspareunia and decreasing libido and responsivity correlated with decreasing estrogen levels.

   - Endostatin (ENST) ENST, a 20-kDa C-terminal fragment cleaved from type XVIII collagen, is a naturally occurring protein that blocks the formation of blood vessels, inhibits EC proliferation, migration and angiogenesis. Furthermore, there is evidence that ENST induces an acute NO release and finally leads to vasodilation and therefore works against endothelial dysfunction.

   However, since there is no data on ENST serum levels in postmenopausal women as well of the effect of Nebivolol on ENST serum levels, we will investigate baseline ENST levels and after 3 month of treatment compared to patients treated with phytohormones.

   - Nebivolol Nebivolol, a ß-blocker of the third generation, has been shown to lower blood pressure with great safety and efficacy in men as well in women and was well tolerated.

   Beneath its specific beta-1-receptor blockade Nebivolol has a NO-releasing effect through a ß3-receptor-agonism. Nebivolol combines a potent ß1-adrenoreceptor-blocking activity (mostly ascribed to its D-enantiomer) with additional vasodilating properties (attributed to its L-enantiomer and also D-enantiomer).

   Nebivolol causes a vasodilatation of the vessels and reduces the progress of atherosclerosis which is a main risk factor for CVD and hypertension.

   The current general guidelines for hypertension recommend treatment with a Thiazide Diuretic as a first line medication in hypertension. In contrary to Diuretics and ACE-blockers - ß-blockers also reduce the heart rate and have positive antagonistic influence on the sympathetic nerve system. The augmentation of the heart rate during the menopause is sensed as a very unpleasant and unbearable situation for most of the postmenopausal women. Thus, the increase in sympathetic nerve activity and clinical symptoms of palpitations or increased heart rate warrant the use of a ß-blocker for the treatment in our cohort.

   Additionally, we hypothesise, that through an improvement of the endothelial function with Nebivolol the number of hot flashes in postmenopausal women can be reduced.

   Recent studies have shown positive effects on the erectile dysfunction in men during treatment with Nebivolol. As the physiologic and embryologic conditions are almost similar in men and women, so we expect similar improving effects on the sexual dysfunction in our female study group.

   Therefore, we want to investigate the effect of Nebivolol on blood pressure, heart rate, hot flashes, sexual function, ENST, testosterone levels in postmenopausal women with menopausal disorders.

   1.2 Rationale of the study

   We want to investigate the effect of Nebivolol in comparison to a phytoestrogen therapy on climacteric disorders as measured by the Menopausal rating scale II (MRS-II). In addition we will investigate the following:

   - the heart rate

   - the number of palpitations

   - the number of hot flushes

   - the sexual function

   - the blood pressure

   - the serum level of Endostatin
   * the serum level of Testosterone in postmenopausal women.

     2 METHODS 2.1 Measurement of the blood pressure Measurement of the blood pressure according to Riva Rocci will be performed at the beginning and after 12 weeks (end of the study). Measurements will be taken in sitting position after five minutes rest. Three consecutive measurements will be taken and the average of these measurements will be recorded.

   2.2 ECG A 12-lead ECG will be written to rule out AV-block and bradycardia (<50/min).

   2.3 Blood parameters

   Prestudy screening:

   - FSH

   - TSH

   - testosterone

   - estrogen

   - DHEA
   * SHBG
   * prolactin
   * BNP
   * hsCRP
   * liver parameters
   * kidney parameters
   * electrolytes
   * blood glucose

   Our patients have to show a blood level of estrogen <20pg/ml and FSH >35 mIU/ml to verify the status of menopause.

   To rule out another endocrine cause of a possible sexual function alteration we check the blood levels of TSH, Prolactin, DHEA (Dehydroepiandrosterone) and SHBG (Sex Hormon Binding Globulin).

   2.4 Analysis of Endostatin Within the routine blood analysis we will also detect the blood level of ENST.

   The RD191076100 Human Endostatin ELISA is a sandwich enzyme immunoassay for the quantitative measurement of endostatin protein in human serum.

   2.5 Female Sexual Function Index We will use the German version of the female sexual function index (FSFI-D) that was validated in 2004. This questionnaire is a proven instrument to evaluate the female sexual function especially in (post)menopausal women.

   We will hand out this questionnaire twice: At the beginning and after our study (12 weeks later). During the completion of the questionnaire by the study participant, a gynecologist will be attendant to help the women to complete the questionnaire.

   This way we want to analyze if the treatment with Nebivolol has an effect on the sexual function of women. We have added the questionnaire to the appendix.

   2.6 Menopausal Rating Scale II We are going to use the Menopause Rating Scale II (MRS II). This self-assessment scale to quantify menopausal symptoms includes 11 questions to evaluate the "quality of life" in our cohort.

   We will hand out this questionnaire twice: At the beginning and after our study (12 weeks later). During the completion of the questionnaire by the study participant, a gynecologist will be attendant to help the women to complete the questionnaire.

   2.7 Hot flashes/palpitations diary At the beginning of our study, the diary will be introduced to the patients by the treating physician. There the number of hot flashes and palpitations per day should be written down. The diary contains 12 pages, one page a week.

   At the beginning we will perform an anamnesis to get informed about the average number of hot flashes and palpitations per day before the medication.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal patients (estrogen <20 pg/ml and FSH >35 mIU/ml)
* The patients are sexually active
* The patients have hot flushes
* The patients have palpitations or extrasystoles

Exclusion Criteria:

Contraindications for a beta-blocker therapy such as:

* Patients with COPD
* Patients with an AV-block
* Patients with a bradycardia (meaning a heart rate <50 beats per minute)
* Patients with hypotension (RR <100/80 mmHg)
* Patients with a PAD (stage III, IV)
* Patients with Asthma
* Patients with Morbus Raynaud
* Patients with a carcinoma
* Patients, who have already been treated because of hypertension
* Patients, who receive hormone replacement therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 Postmenopausal women
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-01

PRIMARY OUTCOMES:
Number of hot flashes/palpitations | 3 Months, 4 appointments
  Number of hot flashes/palpitations during month one and month three compared between nebivolol and phytoestrogens

SECONDARY OUTCOMES:
Hemodynamic changes | 3 Months, 4 appointments
  Measurement of blood pressure and heart rate at baseline and every four weeks.
Sexual function | before and after 3 months of treatment
  Sexual function will be investigated by the Female Sexual Function Index (FSFI-D)
Endostatin | Baseline and after 3 months
  Blood sample of Endostatin will be drawn before and after 3 months of treatment. Endostatin, a cleavage product of collagen XVIII, inhibits angiogenesis. By decreasing neovascualtrization of atherosclerotic plaques, Endostatin might be able to stop the progression of atherosclerosis.
Quality of life | baseline and after 3 months
  Menopause Rating Scale II (MRS II) is a self-assessment scale to quantify menopausal symptoms includes 11 questions to evaluate the "quality of life" in our cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Strametz-Juranek, MD, Principal Investigator — MUV, Department of Internal Medicine II, Division of Cardiology
Locations (1):
- Department of Cardiology, Medical University of Vienna, Vienna, Vienna, Austria